CLINICAL TRIAL: NCT07157527
Title: Impact of Sacubitril/Valsartan Therapy on Left Ventricular Diastolic Function in Patients With Heart Failure With Reduced Ejection Fraction (HFrEF): An Echocardiographic Evaluation
Brief Title: Impact of Sacubitril/Valsartan on LV Diastolic Function in HFrEF
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hebba Awd, resident at the Cardiology Department, Assiut University
Other Study IDs: Sacubitril/Valsartan on LV
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Left Ventricular Diastolic Function
Keywords: Left Ventricular Diastolic Function; Sacubitril; Valsartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receive sacubitril/valsartan as part of guideline-directed medical therapy: Patients receive sacubitril/valsartan as part of guideline-directed medical therapy. Echocardiographic, clinical, ECG, and laboratory evaluations are performed before initiation and after 6 months of continuous ARNI treatment to assess changes in cardiac function and clinical status.

SUMMARY:
This prospective cohort study evaluates the effects of six months of sacubitril/valsartan (ARNI) therapy on left ventricular diastolic function in patients with heart failure with reduced ejection fraction (HFrEF) using transthoracic echocardiography. It aims to correlate echocardiographic parameters with clinical status and systolic function among Egyptian patients treated at two cardiology centers.

DETAILED DESCRIPTION:
Heart failure remains a leading global health issue characterized by high morbidity and mortality, with a pronounced burden in Egypt due to younger patient age and prevalent comorbidities such as diabetes and hypertension. This study addresses the impact of ARNI therapy, which is established for improving systolic outcomes, on diastolic function-an underexplored aspect contributing to symptom severity and prognosis in HFrEF.

Conducted at Assiut General Hospital and Mabarra Hospital cardiology departments, the prospective cohort study enrolls adult patients (≥18 years) with HFrEF (LVEF < 35%) eligible for and initiating sacubitril/valsartan therapy. Transthoracic echocardiography assessments are performed at baseline and after six months of treatment, measuring parameters such as E/A ratio, E/e' ratio, left atrial volume index, deceleration time, and tricuspid regurgitation velocity according to ASE/EACVI guidelines.

The study also integrates clinical evaluations (NYHA class, comorbidities), ECG changes, and laboratory data. Statistical analyses include paired tests to compare changes over time, and correlations between echocardiographic and clinical/laboratory variables. Ethical approval was obtained, and patient confidentiality is assured.

This investigation aims to contribute novel insights into ARNI's effect on diastolic function in a high-risk Egyptian cohort, potentially informing optimized therapy and management of symptomatic heart failure beyond current evidence primarily focused on systolic improvements.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HFrEF (LVEF < 35%)
* Able to tolerate and comply with ARNI therapy
* Patients on Guideline-Directed Medical Therapy (GDMT) for heart failure

Exclusion Criteria:

* Patients with contraindication to ARNI therapy

  * Patients with poor echocardiographic window
  * Patients non-compliant with medication or follow-up
  * Patients with mitral significant lesion or mitral prosthesis.
  * Patients with atrial arrhythmia or on pacemaker

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study enrolls 70 patients characterized by a high prevalence of comorbidities including diabetes mellitus, hypertension, obesity, chronic kidney disease, dyslipidemia, and smoking, reflecting the typical clinical profile of Egyptian HFrEF patients. The median age is younger compared to Western cohorts, with patients presenting advanced heart failure symptoms and poorer functional status. Inclusion criteria require participants to tolerate and comply with ARNI therapy and exclude those with significant mitral valve disease, atrial arrhythmias, pacemakers, or poor echocardiographic windows.
  Comprehensive demographic and clinical data are collected, including sex, NYHA functional class, baseline medications, and heart failure subclassification. This population thus represents a real-world, high-risk group vulnerable to adverse heart failure outcomes, suitable for studying ARNI's effects on diastolic function and overall cardiac remodeling.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Left Ventricular Diastolic Function | Baseline
  Assessment of echocardiographic parameters of diastolic function (E/A ratio)

REFERENCES:
- [Background] Li J, Song Y, Chen F. Evaluating the impact of Sacubitril/valsartan on diastolic function in patients with heart failure: A systematic review and meta-analysis. Medicine (Baltimore). 2024 May 10;103(19):e37965. doi: 10.1097/MD.0000000000037965. PMID 38728489